CLINICAL TRIAL: NCT03028805
Title: Early Patient Identification and Care Pathway for Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial of Informatics Enhanced Hospital Admission
Brief Title: Study of Automated Care Pathway for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: EPICPath
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trend toward increased readmissions in the auto-delivery arm.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ari Hoffman, Assistant Clinical Professor, University of California, San Francisco
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 16-19504
Record Dates: First submitted 2017-01-04; First posted 2017-01-23 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pulmonary Diseases, Obstructive
Keywords: Informatics; COPD; quality improvement
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care and order set A (No Intervention): Usual care. Providers may still search for a COPD order set, and in this arm will see version A, the static list of orders, which is the current state.
- Usual care and order set B (Active Comparator): Usual care in the sense that COPD orders are not automatically included in admission orders despite likelihood of a COPD admission based on the predictive model. However, providers may still search for a COPD order set, and in this arm will see version B, the dynamic list of orders that has been end user tested prior to launch.
  Interventions: Other: Dynamic, end-user order set design
- Automatic inclusion and order set A (Active Comparator): COPD order set is automatically included in admission orders as a static list.
  Interventions: Other: Automatic inclusion of COPD orders in admission orders
- Automatic inclusion and order set B (Active Comparator): COPD order set is automatically included in admission orders as a dynamic and end user tested version.
  Interventions: Other: Automatic inclusion of COPD orders in admission orders; Other: Dynamic, end-user order set design

INTERVENTIONS:
Other: Automatic inclusion of COPD orders in admission orders — Use of real-time data to identify a population of patients with COPD and prompt improved adherence to evidence-based guidelines through the automatic inclusion of a COPD order set in the admission orders.
  Arms: Automatic inclusion and order set A; Automatic inclusion and order set B
Other: Dynamic, end-user order set design — Use of a dynamic order set that has been end-user tested prior to launch rather than designed centrally by a committee to test use of order set components.
  Arms: Automatic inclusion and order set B; Usual care and order set B

SUMMARY:
This is a fully automated randomized trial with two randomization branch-points. The first is inclusion of disease-specific orders in the admission orders based on a predictive model using real-time data. The second is the use of dynamic orders that are end-user tested rather than static orders designed by a committee. The primary hypothesis is that automatic inclusion of disease specific orders with admission orders will improve adherence to guidelines for patients with COPD. The secondary hypothesis is that clinical and operational outcomes will improve, thereby improving value.

DETAILED DESCRIPTION:
This is a single-center, single-blinded, 2x2 factorial randomized controlled trial to test both automated order set inclusion and evidence-based order set design with end user testing on order set use and clinical outcomes for adult patients admitted to the hospital with acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD).

First, the investigators will develop a predictive model to identify patients admitted to the hospital with COPD exacerbations based on retrospective data, but limited to data that is available in real-time at admission.

Second, 1,000 admissions to UCSF Medical Center of adults predicted to have COPD by the predictive algorithm will be prospectively block randomized by encounter to automatic inclusion of a COPD order set in the admission orders or usual care. Providers caring for patients in both arms of the trial can independently search for and use a COPD order set. Any provider using a COPD order set in either arm will also be randomized to see two versions of the order set. The first is a static list of orders, and the second is dynamic, meaning that orders will display only when appropriate. For example, a patient who just had a chest x-ray does not need a routine repeat test. The dynamic order set will show the provider that the x-ray was completed at a specific time and will not display a prompt for a repeat test. Providers can, of course, still order anything they deem clinically appropriate, and may choose to order a repeat x-ray for a patient with a change in clinical status.

The components of the order set are based on international guidelines from the Global Initiative for Chronic Lung Disease (GOLD initiative, a collaboration between the National Heart, Lung, and Blood Institute and the World Health Organization) and a multi-stakeholder working group at UCSF including two hospitalists, two pulmonologists, two transitional care nurse specialists, one advanced practice nurse, one pharmacist, one respiratory therapist, one physical therapist, and one nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or greater admitted to the Hospital Medicine service at UCSF Medical Center who meet criteria as determined by predictive model to be likely admissions for COPD exacerbation.

Exclusion Criteria:

* Patients admitted to other clinical services at UCSF Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Use of evidence-based COPD order set | one year
  Proportion of admissions for COPD exacerbation that use the COPD order set

SECONDARY OUTCOMES:
Average length of stay | one year
Number of inpatient encounters | one year
30-day readmission rates | one year
Mortality | one year
Intubations | one year
Code blue events | one year
ICU admissions | one year
Outpatient utilization | one year
  Encounters for primary care clinic, Pulmonary clinic, Emergency Department or observation during 12 month follow-up
Discharge Disposition | one year
  Proportion of patients discharged to home, home with home health services, or to a facility (includes skilled nursing, acute rehabilitation, sub-acute, long term acute care, and other acute care facilities)
Proportion of enrolled patients billed for COPD related ICD-10 codes for primary or secondary diagnosis. | one year
  ICD-10 codes as described by PRIME program, California's Medicaid 1115 Waiver
Total costs of care | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ari Hoffman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States